CLINICAL TRIAL: NCT03201159
Title: A Pilot, Exploratory Dose Escalating Study on the Safety, Pharmacodynamics and Preliminary Efficacy of VLX103 in the Treatment of Moderate Alcoholic Steatohepatitis
Brief Title: A Pilot, Dose Escalating Study on VLX103 in Moderate Alcoholic Steatohepatitis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug manufacturer ceased operations
Sponsor: Gyongyi Szabo (Other)
Collaborators: The Cleveland Clinic (Other); University of Texas Southwestern Medical Center (Other); University of Louisville (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Gyongyi Szabo, Principal Investigator, University of Massachusetts, Worcester
Organization: University of Massachusetts, Worcester (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: H00011711; VLX103-ASH-16-01 (Other: Verlyx Pharma, Inc); U01AA021893 (NIH)
Record Dates: First submitted 2017-03-24; First posted 2017-06-28 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Hepatic Steatosis
Keywords: ASH
MeSH Terms: conditions — Fatty Liver | interventions — Pentamidine

STUDY DESIGN:
Intervention Model Description: This is a dose escalating Phase Ib study, in which up to 3 doses of VLX103 will be assessed for safety, pharmacodynamics and pharmacokinetics in separate patient cohorts receiving sequentially increasing doses of VLX103. A maximum of 18 well-defined moderate ASH patients will be enrolled and treated in the study, i.e. 6 per dosing cohort.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VLX103 150mg (Experimental): In the first group, 150 mg dosing cohort, one VLX103 tablet will be administered daily for 14 days.
  Interventions: Drug: VLX103
- VLX103 300mg (Experimental): In the second group, 300 mg dosing cohort, two VLX103 tablets will be administered daily for 14 days.
  Interventions: Drug: VLX103
- VLX103 450mg (Experimental): In the third group, 450 mg dosing cohort, three VLX103 tablets will be administered daily for 14 days.
  Interventions: Drug: VLX103

INTERVENTIONS:
Drug: VLX103 — 150mg tablets
  Other Names: Pentamidine Isethionate

SUMMARY:
The study drug (VLX103) is being developed for the treatment of Alcoholic Steatohepatitis and other liver diseases. Alcoholic Steatohepatitis is an inflammatory (associated with irritation, swelling and cell damage) disease that affects the liver. It is associated with heavy and chronic intake of alcohol and presence of fat in the liver. Signs and symptoms often include fever, yellowing of the skin, nausea and impairment of liver function.

The main objective of this study is to evaluate the safety, pharmacodynamics (what the drug does to the body) and pharmacokinetics (how the drug is handled by the human body, like absorption and elimination) of increasing doses of VLX103 in subjects with moderate Alcoholic Steatohepatitis. In other words, we will evaluate how your body tolerates VLX103 at a specific dose and the effects that this VLX103 dose has on your liver and your body in general. The secondary objectives of this study are to evaluate if VLX103 has the potential to treat Alcoholic Steatohepatitis patients, to determine the maximum dose that can be tolerated, and to measure the levels of VLX103 in your blood at different time points during the study.

VLX103 is an experimental drug. Experimental means that the drug has not been approved by the Food and Drug Administration (FDA) for the treatment of Alcoholic Steatohepatitis. The active ingredient in VLX103, pentamidine, is approved for treating parasitic (microorganisms) infections. Pentamidine is currently approved and marketed in about 20 countries, including the United States, for use by injection (administered by a syringe) and by inhalation (administered by a nebulizer) for other health conditions. However, VLX103 is the first oral form of pentamidine being developed, and is administered by mouth as an oral tablet.

DETAILED DESCRIPTION:
This is an open label, multiple cohorts, dose escalation Phase Ib study, in which up to 3 doses of VLX103 will be assessed for safety, pharmacodynamics and pharmacokinetics in well defined moderate ASH patients cohorts receiving increasing doses of VLX103. The overall study design is characteristic for early phase, first in patient clinical evaluation of safety and pharmacodynamics, especially when prudent dose escalation is recommended. A maximum of 18 moderate ASH patients will be enrolled and treated in at least 4 clinical sites throughout the US. The open label nature of the study design will allow to efficiently monitor the safety of VLX103 throughout the trial, and taking rapid decisions about dosing adjustments (dose reduction or discontinuation within each dosing cohort, for each patient).

After an adequate screening period (Day -7 to -1), all eligible patients of the first dosing cohort will receive the initial, low dose of VLX103 150 mg per day (QD) for 14 consecutive days. Subjects will be evaluated only for safety, pharmacodynamics and pharmacokinetics during this period. Pre-established safety criteria will be used to decide upon dose escalation, for each subject. If patients tolerate well VLX103 at 150 mg QD , a second cohort will then receive a 300 mg QD regimen for 14 days. At the end of this period, safety, pharmacodynamics and pharmacokinetics will be assessed as well. The next dose will be 450 mg QD for 14 days, with the same monitoring process. Long term safety will also be assessed, at all 3 doses, at Day 30 and 90 post treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following inclusion criteria:

1. Male and non pregnant female subjects; female subjects must use 2 reliable methods of contraception
2. 18-70 years
3. BMI less than 30 mg/kg2
4. Established diagnosis of Alcoholic Steatohepatitis (ASH), based on at least 2 of the following signs and symptoms should be present: nausea, jaundice, anorexia, right upper quadrant abdominal pain, leukocytosis or hepatomegaly AND
5. Elevation of total bilirubin > 3 mg/dL AND
6. Liver biopsy showing ASH OR ultrasound of liver showing increased echogenicity OR CT scan showing decreased attenuation of liver compared to spleen OR MRI showing fatty liver (decreased signaling intensity on T1 weighted images) History of chronic alcohol consumption, i.e. more than 50 g/day for a minimum of 6 months and at least 2 months before enrolment
7. AST/ALT ratio greater than 1.5
8. MELD score between 12 and 19
9. Signature of a dated Informed Consent Form (ICF) indicating that the subject has been informed of all the relevant aspects of the trial prior to enrolment Willingness and ability to comply with scheduled visits and trial procedures

Exclusion Criteria:

Eligible subjects must not meet any of the following exclusion criteria:

1. Liver disease caused by other etiologies than alcohol (except Hepatitis C and hemochromatosis)
2. Baseline ALT ≥ 200 IU/L
3. Baseline AST ≥ 500 IU/L
4. Signs of systemic infection: fever > 38°C and positive blood or ascites cultures on appropriate antibiotic therapy for ≥ 3 days within 3 days of inclusion
5. Presence of portosystemic encephalopathy at enrolment
6. Presence of cancer at enrolment
7. Presence of uncontrolled diabetes, defined as Hb1Ac ≥ 8.5
8. History of clinically significant hypoglycaemia, with fasting blood glucose < 3 mmol/L within 3 months prior to enrolment
9. Presence of clinically significant renal impairment, defined as serum creatinine ≥ 2.0 x ULN
10. Hypotension with BP < 80/50 mm Hg after volume repletion
11. Current or recent (2 years) history or presence of pancreatitis
12. History of Long QT Syndrome or any significant risk factor for clinically meaningful QT prolongation and Torsades de Pointe.
13. History of significant gastrointestinal surgery that may interfere with the absorption of VLX103
14. Previous treatment with corticosteroids or other immunosuppressive drugs including specific anti-TNF alpha therapy and calcineurin inhibitors within the previous 3 months. Inhaled steroids for asthma are acceptable as long as their use has not been initiated less than 10 days prior to enrolment and their dosing regimen remain stable during the study
15. Concomitant therapy with probiotics, oral neomycin or polymyxin B, rifaximin or other investigational agents or participation in another clinical trial within 3 months of signature of ICF
16. Previous use of pentamidine with treatment discontinuation of less than 12 months prior to study enrolment
17. History of allergy or hypersensitivity to pentamidine
18. Pregnancy or breastfeeding. All female subjects of childbearing potential must have a negative urine pregnancy test prior to first dose of study medication. Breastfeeding is prohibited during the study.
19. Severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgement of the investigator, excess risk associated with trial participation of study drug administration, or which in the judgement of the investigator, would make the subject inappropriate for entry into this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2018-02-27 (Actual); Study Completion 2018-02-27 (Actual)

PRIMARY OUTCOMES:
Frequencies of subjects experiencing at least one adverse event will be displayed by body system and preferred term according to MedDRA terminology | 90 days
  Summary tables will present the number of subjects observed with adverse events and cooresponding percentages. The incidence of adverse events will be summarized by treatment group.
Distribution of laboratory measures over time will be prepared | 90 days
  Listing and summary tables will be prepared for laboratory measures and will be structured to allow review of data by test as the dose is increased

SECONDARY OUTCOMES:
Preliminary efficacy of VLX103 in the target patient population | 7 days and 14 days
  Efficacy as measured by changes in MELD score and serum bilirubin
Maximum Tolerated Dose of VLX103 in moderate ASH patients | 14 days
  determined as the highest safe dose reached according to pre-established safety criteria in the majority of patients
To establish further the hepatoselectivity of VLX103 following up to 14 days of repeated oral administration, through the assessment of systemic drug exposure (serum levels) at selected time points. | 14 days
  assessed by systemic drug levels at selected time points Hepatoselectivity; demonstrated as non significant or absent serum VLX103 levels at Days 7,and 14 and measurable drug concentrations in the liver tissue (if specimens are available).

CONTACTS AND LOCATIONS:
Overall Officials: Gyongyi Szabo, MD, PhD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be filtered through Data Coordinating Center